CLINICAL TRIAL: NCT00765921
Title: A Phase I Single Center Study of Ranibizumab in Combination With Proton Beam Irradiation for Choroidal Melanoma
Brief Title: Ranibizumab in Combination With Proton Beam Irradiation for Choroidal Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-06-040; FVF4384s (Other: Genentech)
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: Choroidal Melanoma
Keywords: glaucoma, neovascular; macular edema; eye enucleation; antibodies, monoclonal; radiation oncology
MeSH Terms: conditions — Uveal Melanoma; Glaucoma, Neovascular; Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.0 mg ranibizumab (Experimental): 1.0 mg intravitreal injection given bi-monthly for 22 months
  Interventions: Drug: ranibizumab
- 0.5 mg ranibizumab (Experimental): 0.5 mg intravitreal injection given bi-monthly for 22 months
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — Ranibizumab dose of 0.5mg or 1.0 mg will be administered intravitreally at the time of surgery for tumor localization and then bimonthly for 22 months (total of 12 injections).
  Other Names: rhuFab; Lucentis

SUMMARY:
The purpose of the study is to investigate the safety and tolerability of the anti-VEGF (vascular endothelial cell growth factor) treatment, ranibizumab, in combination with proton beam irradiation for the treatment of choroidal melanoma by determining the incidence and severity of ocular adverse events. Systemic adverse events will also be evaluated. A secondary objective is to assess the efficacy of ranibizumab in reducing ocular complications that can occur after irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed choroidal melanoma undergoing proton therapy
* Tumors >15 mm in largest diameter and/or >5 mm in height
* Tumors ≤ 15 mm in largest diameter and ≤ 5 mm in height located ≤ 3 mm from optic disc and/or macula, with best-corrected visual acuity 20/100 or better in study eye

Exclusion Criteria:

* History of prior treatment for choroidal melanoma
* Pregnancy or lactation
* Presence of diabetic retinopathy
* History of retinal vascular occlusion or other retinal vascular disease
* Active ocular inflammation or history of uveitis in either eye
* History of uncontrolled glaucoma (defined as intraocular pressure >30mmHg despite treatment with anti-glaucoma medication) or filtering surgery in the study eye
* Previous intravitreal injections of Avastin® in the study eye or in the non-study eye within 30 days.
* Concurrent use of systemic anti-VEGF therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2016-02 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
incidence and severity of ocular adverse events and systemic adverse events | 12 months and 24 months after initial treatment

SECONDARY OUTCOMES:
incidence of radiation-induced complications, vision loss and eye loss | 12 months and 24 months after initial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Kim, M.D., Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye & Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No